CLINICAL TRIAL: NCT05853562
Title: Effects of Structured Exercise Program on Severity of Dizziness, Kinesiophobia, Balance, Fatigue, Quality of Sleep, Activities of Daily Living and Quality Of Life in Bilateral Vestibular Hypofunction
Brief Title: Effects of Structured Exercise Program in Bilateral Vestibular Hypofunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Miray Budak (Other)
Responsible Party: Sponsor-Investigator, Miray Budak, Asst Prof., Istanbul Medipol University Hospital
Organization: Istanbul Medipol University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: BVH_Structured_Exercise
Record Dates: First submitted 2023-04-21; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Bilateral Vestibular Hypofunction
Keywords: Bilateral Vestibular Hypofunction; Dizziness; Kinesiophobia; Balance; Quality of Sleep; Quality of Life; Structured Exercise
MeSH Terms: conditions — Dizziness; Kinesiophobia; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- T0-T1 period (No Intervention): It was a control period. Participants were asked to continue their routine activities for 4 weeks.
- T1-T2 period (structured vestibular rehabilitation program) (Experimental): A structured vestibular rehabilitation program was applied in 50-minute sessions under the supervision of a physiotherapist once a week and as a home exercise program 3 days a week over 4 weeks.
  Interventions: Other: structured vestibular rehabilitation program
- T2-T3 period (Active Comparator): A structured vestibular rehabilitation program was applied in 50-minute sessions under the supervision of a physiotherapist once a week and as a home exercise program 3 days a week over 4 weeks. Afterwards, participants participated in the home program with telerehabilitation for 8 weeks.
  Interventions: Other: structured vestibular rehabilitation program

INTERVENTIONS:
Other: structured vestibular rehabilitation program — The structured Vestibular rehabilitation protocol consisted of a structured vestibular rehabilitation program that included vestibular adaptation exercises, oculomotor exercises, static and dynamic balance exercises, and posture exercises.
  Arms: T1-T2 period (structured vestibular rehabilitation program); T2-T3 period

SUMMARY:
Background: The vestibular rehabilitation is an exercise-based method, aiming to maximize central nervous system(CNS) compensation at vestibular nuclear and other CNS levels for vestibular pathology. A minimal number of studies have documented the impact of Vestibular rehabilitation on the recovery rate of patients with Bilateral Vestibular Hypofunction(BVH).

Objective: The purpose of this study was to investigate the effectiveness of structured vestibular rehabilitation (VR) programs on severity of dizziness, kinesiophobia, balance, fatigue, quality of sleep, activities of daily living( ADL) and quality of life(QoL) in subjects with chronic BVH.

Method: Twenty-five participants diagnosed with BVH were included in the study. A structured VR program was applied in 50-minute sessions once a week and as a home exercise program 3 days a week over 8 weeks. Participants were evaluated for severity of dizziness with the Visual Analog Scale (VAS), for kinesiophobia with the Tampa Scale of Kinesiophobia (TSK), for balance with the Semitandem, tandem, and standing tests, for quality of sleep with the Pittsburgh Sleep Quality Index (PSQI), for ADL with the Vestibular Disorders Activities of Daily Life (VADL), for QoL with Dizziness Handicap Inventory (DHI) and for fatigue with the Fatigue Severity Scale (FSS) at the baseline (T0), at 4th week (T1), 8th week (T2), and 20th week (T3) after study started.

ELIGIBILITY:
Inclusion Criteria:

* Being between 20-80 years old
* Diagnosed with bilateral peripheral vestibular hypofunction by videonystagmography
* Have symptoms for more than three months from onset of illness

Exclusion Criteria:

* having no symptoms of bilateral peripheral vestibular hypofunction
* having Meniere's disease, vestibular migraine and other undulating vestibular disorders, cognitive, visual, neurological or general motor impairment
* having previously received vestibular rehabilitation

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | Change from Baseline Systolic Blood Pressure at 4 / 8 / 12 / 16 weeks
  It is a validated, subjective scale used to measure the intensity or frequency of various symptoms. Scores are based on self-reported measures of symptoms that are recorded with a single handwritten mark placed at one point along the length of a 10-cm line that represents a continuum between the two ends of the scale-"no symptom" on the left end (0 cm) of the scale and the "worst symptom" on the right end of the scale (10 cm). We used this scale to measure the severity of dizziness
Tampa Scale of Kinesiophobia | Change from Baseline Systolic Blood Pressure at 4 / 8 / 12 / 16 weeks
  It is a 17 items self-reporting questionnaire based on evaluation of fear of movement, fear of physical activity, and fear avoidance. The total score of the scale ranges from 17- 68, where 17 means no kinesiophobia, 68 means severe kinesiophobia, and score ± 37 indicates there is kinesiophobia
Semitandem, Tandem, and Standing tests | Change from Baseline Systolic Blood Pressure at 4 / 8 / 12 / 16 weeks
  Semitandem, Tandem, and Standing tests were used to evaluate balance. Semitandem test 30 , Tandem test 30 , Standing tests 30 Equilibrium times (sec) with eyes open-closed were recorded on hard and soft surfaces
Pittsburgh Sleep Quality Index | Change from Baseline Systolic Blood Pressure at 4 / 8 / 12 / 16 weeks
  It is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. The seven component scores consist of subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality
Dizziness Handicap Inventory | Change from Baseline Systolic Blood Pressure at 4 / 8 / 12 / 16 weeks
  It is used to assess the impact of dizziness on quality of life. It consists of 25 clauses which determine the aggravating factors associated with dizziness and shakiness and also the emotional and functional results of vestibular system diseases. The inventory consists of 3 sub-dimensions, intended to determine physical, emotional and functional effects of the vestibular system diseases
Fatigue Severity Scale | Change from Baseline Systolic Blood Pressure at 4 / 8 / 12 / 16 weeks
  It was used to assess fatigue. There are 9 questions in the scale and each question consists of 7 points. An increase in the scale score indicates an increase in the level of fatigue. It detects the state of fatigue in the last month
Vestibular Disorders Activities of Daily Life | Change from Baseline Systolic Blood Pressure at 4 / 8 / 12 / 16 weeks
  This scale is used to determine the degree of independence of patients with vestibular disorders, perceived inadequacies and vestibular complaints in daily activities. The scale consists of 28 items. The subscales are evaluated under three sub-headings as Functional-F- Ambulation-A- and Instrumental-E

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided